CLINICAL TRIAL: NCT03417856
Title: Defining the Skin and Blood Biomarkers of Ichthyosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Galderma R&D (Industry)
Responsible Party: Principal Investigator, Amy Paller, Pediatric Dermatologist, Northwestern University
Other Study IDs: 2014-15801
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Ichthyosis; Netherton Syndrome
Keywords: Ichthyosis; Netherton Syndrome
MeSH Terms: conditions — Ichthyosis; Netherton Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We have retained whole blood and tissue samples (skin and cheek swabs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Healthy subjects with no history of ichthyosis from 1 year to 60 years of age.
- Ichthyosis: Subjects with a diagnosis of Netherton syndrome or ichthyosis from 1 year to 60 years of age.

SUMMARY:
Ichthyosis is a group of genetic skin disorders that present with dry, thickened, scaly, or flaky skin. As of today, there is no cure or treatment. Doctors can only treat the dry skin with different types of emollients to soften the scale. A deeper understanding of this disease is required to develop better treatments. There are different types of cells and cell-produced signals (biomarkers) that are being studied in order to help find these new treatments. Looking at biomarkers has been successful in helping us to understand other skin disorders better. The purpose of this study is to determine which blood and skin biomarkers characterize ichthyosis.

Hypothesis: We predict that the biomarkers correlating with disease activity in Netherton syndrome will be different than the biomarkers found to correlate with the lamellar and other ichthyosis phenotype.

DETAILED DESCRIPTION:
Objectives:

1. To define a panel of skin and blood biomarkers associated with disease activity and pruritus in Netherton syndrome, lamellar ichthyosis, and other ichthyosis subtypes.
2. To determine if blood samples can serve as surrogates for skin immune activation and will correlate with disease severity.
3. To determine FLG, SPINK5, TGM1, or other mutation via buccal/saliva samples in ichthyosis subjects
4. To determine differences in alterations of epidermal lipids and proteins in the outer stratum corneum of epidermis collected from tape strips in patients with ichthyosis compared to the general population. There will also be a difference detected in epidermal lipids from blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Control and ichthyosis subjects may be of either sex and must be between 1-60 years of age at the time of enrollment
* Ichthyosis subjects include individuals with a diagnosis Netherton syndrome, lamellar ichthyosis, or other ichthyosis subtypes
* Ichthyosis subjects should not have administered systemic immunosuppressant therapy in the month before the study
* Ichthyosis subjects should not use topical immunosuppressants in the week before the study
* Ichthyosis subjects should not have applied emollients to the planned biopsy sites within 12 hours before biopsy, but can be applied elsewhere
* Controls may have no inflammatory disease, atopy, or obvious xerosis (urticaria, food allergy, allergic rhinitis or conjunctivitis, asthma)
* Controls for skin sampling may have no observable abnormality in the sampled skin and, to further assure the normality of the "normal" skin edges, must not have evidence of inflammation or epidermal change in the lesion to be surgically removed
* Subjects and guardians of minors must sign the approved IRB consent form(s) prior to initiation of the study protocol

Exclusion Criteria:

* Subjects who are unable to give informed consent or assent
* Subjects who administered anti-inflammatory systemic and topical therapy or emollients that do not comply with inclusion criteria prior to blood and biopsy sampling
* Subjects whose main diagnosis is deemed unsafe by the study investigator for study participation

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 150 subjects (1 year to 60 years of age) with diagnosis of Netherton Syndrome or ichthyosis will be enrolled. Approximately 50 healthy controls will be enrolled. The blood sample, skin biopsy, and buccal/saliva sample may be obtained from the same ichthyosis subject. However there will be separate groups of control patients for the skin biopsies and blood sample studies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cellular infiltrates | One year
  We will examine your skin and blood samples for various immune cells known to be involved in ichthyosis.
Gene expression | One year
  We will examine your skin and blood samples for various genes known to contribute to ichthyosis by analyzing RNA and cytokines.

SECONDARY OUTCOMES:
Correlation of biomarkers to quality of life | One year
  We will analyze the blood and tissue biomarkers to determine whether they are comparable to quality of life and itch (pruritus) measures.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northbrook Lurie Children's Outpatient Clinic, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York